CLINICAL TRIAL: NCT02531737
Title: Multicenter Phase II Trial of Nintedanib (Vargatef®) Plus Docetaxel in Second Line of Treatment in Patients With no Squamous Non Small Cell Lung Cancer Refractory to First Line Chemotherapy
Brief Title: Nintedanib (Vargatef®) Plus Docetaxel in Second Line of Treatment in Patients With Lung Cancer
Acronym: REFRACT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I14041/REFRACT
Record Dates: First submitted 2015-08-18; First posted 2015-08-24 (Estimated); Last update posted 2021-08-10 (Actual); Status verified 2019-07

CONDITIONS: Lung Neoplasms
MeSH Terms: conditions — Lung Neoplasms | interventions — nintedanib; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- traitment (Experimental): Patients will be treated to oral nintedanib (vargatef®) 400 mg/d on days 2 to 21 of a 3-week cycle including docetaxel 75 mg/m2 by intravenous infusion on day 1
  Interventions: Drug: vargatef®; Drug: Docetaxel

INTERVENTIONS:
Drug: vargatef® — Patients will be treated to oral nintedanib (vargatef®) 400 mg/d on days 2 to 21 of a 3-week cycle
  Other Names: Nintedanib
Drug: Docetaxel — Patients will be treated to IV docetaxel 75 mg/m² on day 1 of evry 3-week cycle
  Other Names: Taxotere

SUMMARY:
The purpose of this study is to determine whether nintedanib (vargatef®) combined with docetaxel are effective in second line of treatment in patients with no squamous non small cell lung cancer refractory to first line chemotherapy.

DETAILED DESCRIPTION:
59 Patients with histologically documented stage IV NSCLC no squamous, after failure of first line chemotherapy and refractory (progressive disease during first line chemotherapy), will be enroled to receive docetaxel :75 mg/m² IV day 1 every 3 weeks with nintedanib (vargatef®):200 mg X 2/day per os day2-day21.

Tumor response (according to RECIST) will be assessed via computed tomography or magnetic resonance imaging scan every 6 weeks (evaluation of PFS) following completion of chemotherapy.

Adverse events (AEs) were graded according to the National Cancer Institute Common Toxicity Criteria, version 4.0

Quality of life(EQ5-D ) will be assessed every 6 weeks during chemotherapy. Tolerability will be assessed at each visit based on Common Terminology Criteria for Adverse Events (CTCAE), v4.0 criteria.

Total study duration per patient: approximately 12 months .

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed non-squamous NSCLC,
* Metastatic NSCLC of stage IV (according to American Joint Committee on Cancers) or recurrent NSCLC)
* Patients without activating epidermal growth factor receptor (EGFR) mutation
* Patients without anaplastic lymphoma kinase (ALK) rearrangement
* Patients must have measurable lesion by RECIST 1.1
* Refractory disease defined by documented progression during the first-line chemotherapy based on a platinum doublet and third-generation drug (four or less cycles) according to RECIST V.1.1
* Age ≥18 years and < 75 years
* Performance status (PS) 0-1
* Life expectancy of more than 12 weeks.
* No history of other malignancy within the last 5 years, except for adequately treated carcinoma in situ of the cervix or basal cell or spinocellular carcinoma of the skin.
* Adequate organ function, evidenced by the following laboratory results within 3 weeks prior to randomization: Normal hepatic function: bilirubin < 1.5 x N, ALT (alanine transaminase) and AST (aspartate aminotransferase ) < 2.5 x N or <5 x N in case of liver metastasis
* Normal renal function (calculated creatinine clearance ≥ 45 mL/min).
* Normal Calcemia
* Normal haematological function (polynuclear neutrophils > 1.5 G/l, platelets > 100 G/l).
* Anticoagulation with a vitamin K antagonist and low-molecular-weight heparin (LMWH) is authorized.
* Antiplatelet treatment (aspirin authorized if < 325 mg/d)
* Treatment with dipyridamole, ticlopidine, clopidogrel is not authorized
* Women of child bearing potential must use double effective contraception.
* Men might be surgically sterile or accept to use an effective contraceptive procedure during and until 6 months after the treatment.
* Written informed consent to participate in the study.

Exclusion Criteria:

* Known hypersensitivity to the trial drugs (nintedanib (vargatef®), docetaxel), peanut, soya, to their excipients
* Controlled disease after first line treatment
* Contra indication to the use of the backbone treatment
* Patients who were withdrawn from first line treatment due to toxicity without documented disease progression or who received placebo (in the context of a clinical trial) as prior treatment are not eligible.
* Previous treatment with docetaxel
* Small-cell lung cancer, bronchioloalveolar cancer, neuroendocrine cancer.
* Previous therapy with vascular endothelial growth factor (VEGF) inhibitors except bevacizumab
* Centrally located tumour with radiographic evidence of local invasion of local blood vessels
* Radiographic evidence of cavitary or necrotic tumours at screening
* Chemo-, hormone-, radio-(except for brain and extremities) or immunotherapy or therapy with monoclonal antibodies or small tyrosine kinase inhibitors within the past 4 weeks prior to treatment with the trial drug.
* Toxicity non resolute due to prior treatment > grade I (except alopecia).
* Radiotherapy (except extremities) within the past 3 months prior to baseline imaging
* Persistence of clinically relevant therapy related toxicity from previous radiotherapy
* Active brain metastases (e.g. stable for <4 weeks, no adequate previous treatment with radiotherapy, symptomatic, requiring treatment with anti-convulsants; dexamethasone therapy will be allowed if administered as stable dose for at least one month before inclusion).
* Uncontrolled arterial hypertension.
* Concurrent radiotherapy, except for palliative bone irradiation.
* Other concurrent severe illnesses (congestive heart failure, unstable angina, significant arrhythmia or myocardial infarction less than 12 months before study entry).
* Stroke less than 6 months before study entry.
* Psychiatric or neurological disorders preventing the patient from understanding the nature of the trial
* Grade >=1 peripheral neuropathy
* Uncontrolled infection.
* Caval syndrome
* Other organic disorders preventing inclusion in the trial
* Malabsorption syndrome
* Pregnancy and breast-feeding
* Surgery less than two months before study entry.
* Follow-up not feasible.
* Incarcerated and institutionalized

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2020-09-26 (Actual); Study Completion 2020-09-26 (Actual)

PRIMARY OUTCOMES:
median progression free survival | 12 weeks

SECONDARY OUTCOMES:
median progression free survival | 12 month
Toxicity (NCIC-CTC version 4.0 criteria) | Every 3 weeks during treatment up to 12 months from inclusion
Quality of life (EQ5-D questionnaire) | every 6 weeks up to 12 months from inlcusion
Response rate | 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Alain Vergnenegre, MD, Principal Investigator — CHU LImoges
Locations (11):
- France (11):
  - CH de Beauvais, Beauvais
  - CHU Brest, Brest
  - Service de Pneumologie, Créteil
  - Service de Pneumologie, Gap
  - CHU de Limoges, Limoges
  - CH de Bretagne Sud, Lorient
  - Centre Hospitalier F. Quesnay, Mantes-la-Jolie
  - AP-HM, Marseille
  - Institut Paoli-Calmettes, Marseille
  - Instiut de Cancérologie, Saint-Etienne
  - Service de Pneumologie, Villefranche